CLINICAL TRIAL: NCT06978478
Title: An Imaging Feasibility Study in Oestrogen Receptor Negative MEtastatic Breast Cancer by Targeting Integrin Alpha -v Beta 6
Brief Title: An Imaging Study in ER Negative Breast Cancer by Targeting αvβ6
Acronym: IMETAB6
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: EDGE Suspended 27/09/2022
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 010954QM
Record Dates: First submitted 2017-08-29; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): Pilot study: All registered patients will undergo 2 CT PET scans.
  Interventions: Procedure: Unlabelled PET CT Scan; Procedure: Labelled PET CT Scan

INTERVENTIONS:
Procedure: Unlabelled PET CT Scan — [18F]-FDG-PET CT
Procedure: Labelled PET CT Scan — [18F]-FBA-A20FMDV2 -PET CT

SUMMARY:
This is a multicentre, pilot study that aims to determine the feasibility of [18F]-FBA-A20FMDV2-PET CT scans to detect levels of αvβ6 in patients with ER-ve αvβ6-positive metastatic or locally advanced breast cancer. A combination of factors will be used to determine the feasibility of [18F]-FBA-A20FMDV2-PET CT imaging including visual adequacy of the PET CT image, adequate signal to noise ratio and the ability to evaluate the image differential between the metastatic lesion(s) and normal tissue.

DETAILED DESCRIPTION:
Integrin alpha v beta six (αvβ6) is present in increased amounts on a number of cancer cells and is known to play a prominent role in cancer development and spread. FBA-A20FMDV2 is a substance that sticks to αvβ6. It may therefore be possible to identify and measure the amount of αvβ6 in tumours by attaching a small amount of radioactivity to FBAA20FMDV2 and carrying out a scan called a PET scan. FBA-A20FMDV2 attached to radioactivity is known as [18F]-FBAA20FMDV2 or a radiotracer, where very small amount of tracer doses are given to man.

Such scans have been carried out in healthy volunteers and patients with a lung condition to assess radiotracer safety and specificity. IMETAB6 will help to find out how [18F]-FBA-A20FMDV2 is taken up in tumours in breast cancer patients where their cancer has spread (metastasised) to other parts of the body. This information will be used to develop the ideal imaging method for cancer patients where their disease has metastasised.

20 women with hormone (oestrogen) receptor (ER)-negative breast cancer whose tumours contain αvβ6, measure

≥1cm in diameter, and whose cancer has metastasised, will be on the study for 4 weeks. These women will give blood samples and undergo one [18F]-FBA-A20FMDV2-PET scan, and one 'control' scan without FBA-A20FMDV2 (an FDG-PET scan) for comparison, to see if tumours containing αvβ6 can be detected. Participants will be called within 3 days following their [18F]-FBA-A20FMDV2-PET scan to check their wellbeing. All patients will be recruited from Barts Health NHS Trust oncology clinics, where they will undergo an [18F]-FDG-PETCT scan. They will then undergo the [18F]-FBA-A20FMDV2-PET scan at Imanova Centre for Imaging Sciences. αvβ6 levels will be measured on patient tumour samples as part of their normal clinical care and a small sample (biopsy) of their metastasis will be analysed for αvβ6.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give written informed consent prior to admission to this study.
2. Female aged ≥18 years.
3. ECOG performance status of 0-2.
4. Histologically confirmed ER-ve metastatic or locally advanced breast cancer (latest available sample). ER-ve status defined as <1% of tumour cells positive for ER on IHC or IHC score (Allred) ≤2. Any HER2 status is acceptable.
5. At least one metastatic tumour site measuring ≥1cm in the longest diameter (except lymph nodes which must have a short axis of ≥1.5cm) as assessed by clinical imaging or by physical clinical evaluation.
6. Biopsiable metastatic or locally advanced tumour sites, if a FFPE sample of current metastatic sites is not available. If an FFPE sample from the current metastatic sites is not available then patients must be willing to undergo an US or CT guided biopsy.
7. Available FFPE tumour sample of the primary tumour prior to study entry for central assessment.
8. Known αvβ6 status on primary or metastatic tumour (latest available) as defined by IHC.
9. Patient must be progressing on current anti-cancer treatment (non-responder).
10. Haematologic indices (FBC, WBC, ANC, platelets count and haemoglobin) and biochemical indices (sodium, potassium, chloride, urea, creatinine, total protein, albumin, total bilirubin, ALP and AST) within local institutional limits.
11. Negative serum or urine pregnancy test for female patients of childbearing potential prior to study entry . Female patients of childbearing potential must agree to use adequate contraception as described in the protocol from the day of the scan and until 4 weeks after the last scan.

Exclusion Criteria:

1. Breast-feeding female patients.
2. Previous or current exposure to animals that may harbour the foot and mouth disease virus FMDV2
3. Previous long-term (≥ 3 months) residence in a country where FMDV2 is endemic (such as certain areas of Africa, Asia and South America).
4. Planned to receive further anti-cancer treatment while on study.
5. Subject feels unable to lie flat and still on their back for a period of up to 95 minutes in the PET/CT scanner.
6. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of the tracer, may affect the interpretation of the results, render the patient at high risk from treatment complications or interferes with obtaining informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female only
Enrollment: 0 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Uptake of [18F]FBA-A20FMDV2 in tumours expressed as standardised uptake value | Through study completion of 4 weeks - Study withdrawn and no further information
  Imaging results will be continuously assessed before proceeding to the next patient and the timing of the radiotracer administration in relation to the scan start will be varied to optimise image acquisition.

SECONDARY OUTCOMES:
Concordance between [18F]-FBA-A20FMDV2-PET CT scans and [18F]-FDG-PET CT scans. | Through study completion of 4 weeks - Study withdrawn and no further information]
  Study withdrawn - no further information
Correlate [18F]-FBA-A20FMDV2-PET CT uptake measures with standard IHC expression in metastatic tumour samples. | Through study completion of 4 weeks - Study withdrawn and no further information]
  Study withdrawn - no further information
Change in αvβ6 expression levels in primary and metastatic tumour samples by IHC. | Through study completion of 4 weeks - Study withdrawn and no further information]
  Study withdrawn - no further information

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, Principal Investigator — Queen Mary University of London; John Marshall, Principal Investigator — Queen Mary University of London
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No